CLINICAL TRIAL: NCT03080493
Title: Gabapentin for Pain Control After Osmotic Dilator Insertion and Prior to D&E Procedure: a Randomized Controlled Trial
Acronym: GABA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 987072
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Abortion, Induced; Cervical Preparation; Pain
Keywords: Abortion; Osmotic dilators; Gabapentin; Text message
MeSH Terms: conditions — Pain | interventions — Gabapentin; Carboxymethylcellulose Sodium; Acetaminophen; Codeine; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled trial, stratified block randomization based on prior vaginal parity (vaginal parity - yes or no). Goal of even distribution of prior vaginal parity between gabapentin and placebo groups as may impact osmotic dilator pain experience
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin 600 mg PO - first dose in clinic prior to osmotic dilator placement, second dose 8 hours later (at home)
  Will receive standard regimen of acetaminophen/codeine and ibuprofen to take as needed for pain overnight
  Interventions: Drug: Gabapentin 600mg; Drug: acetaminophen/codeine and ibuprofen
- Placebo oral capsule (Placebo Comparator): Matched placebo
  Will receive standard regimen of acetaminophen/codeine and ibuprofen to take as needed for pain overnight
  Interventions: Drug: Placebo oral capsule; Drug: acetaminophen/codeine and ibuprofen

INTERVENTIONS:
Drug: Gabapentin 600mg — Gabapentin 600 mg PO (two total doses, thereby lasting duration while osmotic dilators are in place)
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo oral capsule — Packaged identical to gabapentin dosing
  Other Names: Carboxymethyl cellulose
  Arms: Placebo oral capsule
Drug: acetaminophen/codeine and ibuprofen — Over the counter analgesic medications
  Other Names: Tylenol-Codeine No. 3; Advil

SUMMARY:
Women having abortion procedures between 15 weeks 0 days and 23 weeks 6 days gestational age on the day of their procedure commonly have dilators placed in their cervix overnight before the abortion procedure. The dilators are put in during a pelvic exam in the clinic and after women go home they expand slowly overnight to open the cervix before the abortion procedure the next day. This can be a painful experience and health care providers often give women different kinds of pain medicine to help them.

The investigators are interested in whether a medicine called gabapentin, which is a non-narcotic medicine, could help. Gabapentin is approved by the U.S. Food and Drug Administration (FDA) for prevention of seizures and for treating nerve pain and doctors are also using it to decrease pain for people having surgical procedures.

The main goals of our study are to learn about:

1. Women's pain experience with dilators in their cervix overnight before the abortion procedure
2. How well gabapentin works to decrease women's pain while they have the dilators in their cervix

Women who enroll in the study will get a dose of either gabapentin or placebo (a pill with no medicine in it) before their dilators are placed in the clinic. The medication they get (gabapentin or placebo) will be chosen by chance, like flipping a coin. Neither the women in the study nor the doctors giving them the medication will know which medication they receive so the investigators can learn about their pain without being influenced by knowing which medication they take. Doctors will be able to find out which medication women got if there is an emergency or if it changes their medical care.

The investigators will communicate with women in real time overnight by text messaging to see how much pain they are having in the moment and how much pain medicine they are taking.

The investigators hypothesize that women who receive gabapentin will have a smaller increase in their pain with the dilators than women who receive placebo (a pill with no medicine in it).

The investigators' findings will help doctors understand women's pain experience with dilators better and possibly provide a new way of treating pain with gabapentin.

DETAILED DESCRIPTION:
The investigators have planned a double-blind randomized controlled trial of repeated doses of gabapentin compared to placebo for pain management during the time after dilator insertion and prior to D&E the subsequent day.

* Participants will receive gabapentin 600 mg or placebo prior to dilator insertion
* Pain scores will be measured via numeric rating scale (NRS) at baseline and 5 minutes after last dilator insertion while the participant is in clinic
* Additional pain scores, side effects (specifically dizziness and sedation), and additional analgesic use will be obtained by text message while the patient is home at 2 hours, 4 hours, and 8 hours after time of dilator insertion
* Subjects will take a second dose of study drug (either gabapentin 600 mg or placebo, concordant with their initial medication) at 8 hours after their first dose
* Final pain score, side effect, and analgesic use assessment will occur upon presentation to the pre-operative are for D&E the subsequent day

There will be no change in standard insertion of osmotic dilators (hygroscopic dilators only with Lidocaine 20mL cervical anesthesia), or provision of home analgesic medications (ibuprofen and acetaminophen with codeine in our practice).

The investigators hypothesize that women who receive gabapentin will report a smaller increase in pain from baseline at 8 hours after dilator placement compared to women receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* 15 weeks 0 days gestational age - 23 weeks 5 days gestational age at time of dilator insertion
* Able to read and write in English
* Active cell phone with text messaging capability
* Ride home from dilator insertion clinic appointment

Exclusion Criteria:

* Current use of gabapentin or pregabalin
* Allergy to gabapentin, acetaminophen, codeine, or ibuprofen
* Self reported renal disease (severe impaired renal function)
* Self reported current or chronic narcotic use (typical daily use)
* Women with any issue that, in the opinion of the investigator, would interfere with study participation or generating accurate study data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Schimmoeller, MD, MPH, MA, Principal Investigator — University of California, Davis; Mitchell Creinin, MD, Study Director — University of California, Davis
Locations (1):
- University of California Davis Health System, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan PZ, Butler PM, Kurowski D, Perloff MD. Beyond neuropathic pain: gabapentin use in cancer pain and perioperative pain. Clin J Pain. 2014 Jul;30(7):613-29. doi: 10.1097/AJP.0000000000000014. PMID 24281281
- [Background] Rose MA, Kam PC. Gabapentin: pharmacology and its use in pain management. Anaesthesia. 2002 May;57(5):451-62. doi: 10.1046/j.0003-2409.2001.02399.x. PMID 11966555
- [Background] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin 600 mg PO - first dose in clinic prior to osmotic dilator placement, second dose 8 hours later (at home)
  Will receive standard regimen of acetaminophen/codeine and ibuprofen to take as needed for pain overnight
  Gabapentin 600mg: Gabapentin 600 mg PO (two total doses, thereby lasting duration while osmotic dilators are in place)
  acetaminophen/codeine and ibuprofen: Over the counter analgesic medications
- Placebo Oral Capsule: Matched placebo
  Will receive standard regimen of acetaminophen/codeine and ibuprofen to take as needed for pain overnight
  Placebo oral capsule: Packaged identical to gabapentin dosing
  acetaminophen/codeine and ibuprofen: Over the counter analgesic medications
Period: Overall Study
Arm/Group | Gabapentin | Placebo Oral Capsule
Started | 61 | 60
Completed | 60 | 58
Not Completed | 1 | 2
Not completed — Did not provide NRS pain results | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Randomization error (parity group) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo Oral Capsule | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.6) | 27.2 (6.1) | 26.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 42 | 85
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 23 | 34 | 57
  Race: Black | 11 | 11 | 22
  Race: Asian | 7 | 3 | 10
  Race: Mixed | 14 | 5 | 19
  Race: Other | 4 | 2 | 6
  Race: Declined | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118
Reasons for abortion [Count of Participants; unit: Participants]
  Unwanted pregnancy | 53 | 51 | 104
  Fetal anomalies | 7 | 7 | 14
Education [Count of Participants; unit: Participants]
  Not completed high school | 6 | 4 | 10
  High school or equivalent | 30 | 15 | 45
  Some college | 16 | 32 | 48
  College or higher | 8 | 6 | 14
  Declined | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in NRS Pain Score at 8 Hours After Dilator Insertion
Description: Pain score based on numeric rating scale (NRS [0 lowest value to 10 highest value, in which 0 is the lowest amount of pain and 10 is the highest amount of pain]); Baseline obtained prior to study drug ingestion/dilator insertion. NRS pain score obtained via text message.
Time Frame: 8 hours after insertion of last osmotic dilator
Population: Women who responded with pain scores by text using Numeric Rating Scale
Measure: Median (Full Range); unit: Numeric rating scale pain score change
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 58 | 52
Numeric rating scale pain score change | 2 [-3 to 8] | 2.5 [-5 to 10]

2. Secondary Outcome: Mean Change From Baseline in NRS Pain Score at 5 Minutes After Last Dilator Insertion
Description: Pain score based on numeric rating scale (NRS [0 lowest value to 10 highest value, in which 0 is the lowest amount of pain and 10 is the highest amount of pain]); Baseline obtained prior to study drug ingestion/dilator insertion. NRS pain score obtained in person before subject leaves clinic appointment.
Time Frame: 5 minutes after insertion of last osmotic dilator
Population: Women who provided Numeric rating scale pain score
Measure: Median (Full Range); unit: Numeric rating scale pain score change
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 60 | 58
Numeric rating scale pain score change | 1 [-6 to 10] | 2 [-5 to 8]

3. Secondary Outcome: Mean Change From Baseline in NRS Pain Score at 2 Hours After Dilator Insertion
Description: as for outcome 1
Time Frame: 2 hours after insertion of last osmotic dilator
Population: Women who responded by text with numeric pain scale score
Measure: Median (Full Range); unit: Numeric rating scale pain score change
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 54 | 54
Numeric rating scale pain score change | 3.5 [-8 to 9] | 4 [-2 to 10]

4. Secondary Outcome: Mean Change From Baseline in NRS Pain Score at 4 Hours After Dilator Insertion
Description: as for outcome 1
Time Frame: 4 hours after insertion of last osmotic dilator
Population: Women who responded by text with numeric pain scale score
Measure: Mean (Full Range); unit: Numeric rating scale pain score change
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 56 | 50
Numeric rating scale pain score change | 3 [-8 to 9] | 3.5 [-3 to 10]

5. Secondary Outcome: Mean Change From Baseline in NRS Pain Score at Time of Presentation for D&E Procedure (Day Following Dilator Insertion)
Description: Pain score based on numeric rating scale (NRS [0 lowest value to 10 highest value, in which 0 is the lowest amount of pain and 10 is the highest amount of pain]); Baseline obtained prior to study drug ingestion/dilator insertion. NRS pain score obtained in person upon presentation for D&E procedure.
Time Frame: Time of presentation for D&E (day after dilator insertion)
Population: Women who provided numeric pain scale scores
Measure: Median (Full Range); unit: Numeric rating scale pain score change
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 60 | 58
Numeric rating scale pain score change | 0.5 [-8 to 7] | 1 [-2 to 9]

6. Secondary Outcome: Number of Participants Using Narcotic Pain Medication (Acetaminophen/Codeine)
Description: Subject account of how many used acetaminophen/codeine (standard medications given for supplement NSAID as needed after dilator insertion)
Time Frame: Collected between each subject contact (2 hours, 4 hours, 8 hours after dilator insertion and at time of presentation for D&E procedure)
Population: Any use of narcotics
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 60 | 58
Participants | 35 | 40

ADVERSE EVENTS:
Time Frame: One day (from treatment initiation until procedure the following day
Description: Only adverse events collected were specific to the intervention: dizziness and tiredness
Arm/Group | Gabapentin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 57/60 | 51/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Gabapentin (N=60) | Placebo Oral Capsule (N=58)
Dizziness at baseline (Nervous system disorders) | 1 (1) | 0 (0) — Dizziness
Dizziness at 5 minutes after dilator placement (Nervous system disorders) | 21 (21) | 15 (15) — Dizziness
Dizzines at 2 hours after dilator placement (Nervous system disorders) | 29/53 (29) | 11/53 (11) — Dizziness
Dizziness at 4 hours after dilator placement (Nervous system disorders) | 22/55 (22) | 5/50 (5) — Dizziness
Dizziness at 8 hours after dilator placement (Nervous system disorders) | 15/57 (15) | 3/52 (3) — Dizziness
Dizziness at 18-24 hours after dilator placement (Nervous system disorders) | 3 (3) | 4 (4) — Dizziness
Tiredness at baseline (General disorders) | 7 (7) | 4 (4) — Tiredness
Tiredness at 5 minutes after dilator placement (General disorders) | 7 (7) | 12 (12) — Tiredness
Tiredness at 2 hours after dilator placement (General disorders) | 34/54 (34) | 17/54 (17) — Tiredness
Tiredness at 4 hours after dilator placement (General disorders) | 37/54 (37) | 18/51 (18) — Tiredness
Tiredness at 8 hours after dilator placement (General disorders) | 22/57 (22) | 17/51 (17) — Tiredness
Tiredness at 18-24 hours after dilator placment (General disorders) | 18 (18) | 22 (22) — Tiredness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03080493/Prot_SAP_000.pdf